CLINICAL TRIAL: NCT02270697
Title: Evaluation of an Oligonucleotide Array for Rapid Identification of Dermatophytes in Clinical Specimens
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Tsung Chain Chang, Professor, National Cheng-Kung University Hospital
Other Study IDs: A-ER-101-336
Record Dates: First submitted 2014-10-16; First posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Tinea Unguium; Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — * Nail Samples
  * Scrap Samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Regular Diagnosis: Difficult in regular diagnosis specimens, assistance with array.
  Interventions: Device: Array

INTERVENTIONS:
Device: Array — Applications of oligonucleotide array in diagnosis.

SUMMARY:
The nail specimens from patients with suspect onychomycosis were analyzed. Samples were collected as part of standard patient care from the Department of Dermatology, National Cheng Kung University Hospital (NCKUH, a tertiary referral hospital), Tainan, Taiwan. Comparing the array results with the regular methods by sensitivity, specificity, NPV and PPV.

DETAILED DESCRIPTION:
The nail specimens from patients with suspect onychomycosis were analyzed.

Collection:

Samples were collected as part of standard patient care from the Department of Dermatology, National Cheng Kung University Hospital (NCKUH, a tertiary referral hospital), Tainan, Taiwan.

Nail samples were collected as subungual scrapings, clippings, or curettings. Samples were immediately transported in sterile Eppendorf tubes at room temperature to the laboratory of Department of Dermatology, NCKUH, for KOH stain and routine fungal cultures.

Sample Prepare:

Each sample was cut into small pieces with a surgical blade and homogenization by 2-ml glass homogenizer. The suspension treated by lyticase at 37°C for 30 min and extracted DNA with Blood & Tissue genomic DNA kit.PCR program and array hybirdization same with previous study.

Analysis:

If the results between array and culture method, discrepant analysis with re-sequencing, KOH mount and the patient's outcome of after antifungal treatment. The performance evaluation of the array and culture methods with Sensitivity, specificity, positive (PPV) and negative predictive value (NPV) were calculated after discrepant analysis. Significant difference was estimated by Fisher's exact test.

ELIGIBILITY:
Inclusion Criteria:

* Atypically results by culture and microscopy
* Suspect tinea infection

Exclusion Criteria:

* Lost follow
* Not tinea unguium

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subject were suspect onychomycosis and treatment at National Cheng Kung University Hospital.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Oligonucleotide Array Detection Resluts | 1 weeks
  The species of pathogen provide by array method.

CONTACTS AND LOCATIONS:
Overall Officials: Tsung Chain Chang, PhD, Principal Investigator — National Cheng Kung University